CLINICAL TRIAL: NCT00833976
Title: Omega-3 Fatty Acids (Lovaza) for Second Generation Antipsychotic-Associated Hypertriglyceridemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Marlene P. Freeman, MD, Director of Clinical Services, MGH Center for Women's Mental Health, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-P-002219
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: High Triglycerides; Hypercholesterolemia; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
MeSH Terms: conditions — Hypertriglyceridemia; Hypercholesterolemia; Schizophrenia; Psychotic Disorders; Bipolar Disorder | interventions — Omacor; Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open-label Lovaza (omega-3 fatty acids) (Experimental): 4g per day (4g once a day or 2g two times a day) for 16 weeks
  Interventions: Drug: Lovaza

INTERVENTIONS:
Drug: Lovaza — 4 grams per day
  Other Names: Omega 3 Fatty Acids

SUMMARY:
This is an open-label pilot study of omega-3 fatty acids (Lovaza) for hypertriglyceridemia in subjects who have been on an atypical (second-generation) antipsychotic medication. The investigators hypotheses are that patients who receive Lovaza will experience a significant decrease in triglycerides from baseline. Secondary hypotheses include: Patients will experience a significant decrease in total cholesterol, and Lovaza will be well tolerated.

DETAILED DESCRIPTION:
This is an open-label pilot study of omega-3 fatty acids (Lovaza) for hypertriglyceridemia in subjects who have been on an atypical (second generation) antipsychotic medication. Eligible subjects include men and women, ages 18-75, who have been taking an atypical antipsychotic for at least three months prior to enrollment. Atypical antipsychotics include: clozapine (Clozaril), olanzapine (Zyprexa), risperidone (Risperdal), aripiprazole (Abilify), ziprasidone (Geodon), quetiapine (Seroquel), paliperidone (Invega), asenapine (Saphris), iloperidone (Fanapt), and lurasidone (Latuda). Eligible subjects must also have serum triglycerides >200 mg/dl or high cholesterol >250 mg/dl at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients, 18-75 years of age.
2. Serum triglycerides >200 mg/dl or high cholesterol >250 mg/dl
3. Current use of an atypical (second-generation) antipsychotic medication - including clozapine (Clozaril), olanzapine (Zyprexa), risperidone (Risperdal), aripiprazole (Abilify), ziprasidone (Geodon), quetiapine (Seroquel), paliperidone (Invega) - for at least three months

Exclusion Criteria:

1. Current use of triglyceride or cholesterol-lowering medication other than a statin
2. Current use of omega-3 fatty acid supplement
3. Intake of fish more than twice per week
4. Currently pregnant, or breastfeeding
5. Known hypersensitivity or allergy to omega-3 fatty acids (or any fish allergies)
6. Current use of anticoagulant medication, except for 1 baby aspirin/day - 81mg (coumadin, heparin, Plavix. etc).
7. Consumption of alcohol greater than two drinks per day or active substance abuse
8. Any medical condition that would make participation in the study unsafe, as determined by investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene P Freeman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Massachusetts General Hospital's Center for Women's Mental Health — http://www.womensmentalhealth.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-label Lovaza (Omega-3 Fatty Acids)
Started | 65
Completed | 14
Not Completed | 51
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 4
Not completed — Did not meet eligibility criteria | 41
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Lovaza (Omega-3 Fatty Acids)
Number analyzed (Participants) | 65
Age, Continuous [Median (Standard Deviation); unit: years] | 48 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Change in Triglycerides From Baseline to 16 Weeks
Time Frame: 16 weeks
Population: Although only 14 participants completed the triall, 16 were included in the analyzable population. The 2 participants who are analyzable but not completers were lost to follow-up. They were included in the analysis since they still had 2 measurements time points. These 16 participants all had adherence values, as determined by pill count, of ≥75%
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open-label Lovaza (Omega-3 Fatty Acids)
Number analyzed (Participants) | 16
mg/dL | -54.13 (83.44)

2. Secondary Outcome: Change in Total Cholesterol From Baseline to 16 Weeks
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open-label Lovaza (Omega-3 Fatty Acids)
Number analyzed (Participants) | 16
mg/dL | -1.75 (29.40)

3. Secondary Outcome: Tolerability of Omega-3 Fatty Acid Capsules (Lovaza)
Description: At each of the visits, participants completed a questionnaire to determine tolerability of the omega-3 fatty acid capsules (Lovaza).
Time Frame: 16 weeks
Population: All participants who took at least one dose of the study medication were included in the analyzable population.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Lovaza (Omega-3 Fatty Acids)
Number analyzed (Participants) | 23
Participants
  non-tolerable | 1
  tolerable | 22

ADVERSE EVENTS:
Arm/Group | Open-label Lovaza (Omega-3 Fatty Acids)
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 13/65
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Lovaza (Omega-3 Fatty Acids) (N=65)
Nausea (Gastrointestinal disorders) | 4 (5)
Abnormal potassium levels (Renal and urinary disorders) | 2 (2)
Abnormal levels of sodium (Renal and urinary disorders) | 1 (1)
Dehydration (Renal and urinary disorders) | 1 (1)
Unpleasant taste (Gastrointestinal disorders) | 2 (2)
Chest pain (Cardiac disorders) | 1 (1)
Compulsive eating (Psychiatric disorders) | 1 (1)
Gassy (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No